CLINICAL TRIAL: NCT00109460
Title: Tobacco Cessation Clinical Field Study for Adults in Alcohol Abuse Recovery
Brief Title: Tobacco Cessation Field Study for Adults in Recovery - 1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Inflexxion, Inc. (Industry)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Model: Crossover | Masking: Single
Other Study IDs: NIDA-80460-1; R44DA080460 (NIH)
Record Dates: First submitted 2005-04-27; First posted 2005-04-28 (Estimated); Last update posted 2015-05-13 (Estimated); Status verified 2015-05

CONDITIONS: Tobacco Use Disorder
Keywords: Tobacco
MeSH Terms: conditions — Tobacco Use Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Behavioral: Tobacco Use Disorder

SUMMARY:
The project's aim is to provide a targeted, computer-administered intervention to facilitate tobacco cessation for clients in alcohol treatment. The main focus of "On the Air: A tobacco cessation program for adults in alcohol recovery" is to reduce tobacco use of clients in alcohol treatment. The program will be offered through inpatient, residential, and outpatient treatment programs to help those struggling with alcohol addiction to understand, reduce, and stop tobacco use. Clients will develop a personalized tobacco cessation plan relevant to their readiness to quit tobacco use. Based on the metaphor of a television network, this tobacco cessation program contains information on personal risks, peer stories, cravings and withdrawal, a variety of interactive activities and tools, and also motivational feedback and tips to assist in the quitting process. Phase I was a proof of concept phase, in which we delivered a prototype CD-ROM on tobacco cessation. Phase II will involve completing the development of a functional CD-ROM tool which will be subjected to a clinical field trial with a group of adults (n=196) in treatment facilities for alcohol recovery. The clinical field study will involve finalizing the content, interface, and interactive features of the CD-ROM. We will also gather satisfaction data from both clients and counselors in the various treatment facilities.

ELIGIBILITY:
Inclusion Criteria:

* Carry a primary DSM-IV diagnosis of alcohol abuse or dependence
* Smoke at least one cigarette a day
* Be willing to sign informed consent and undergo initial assessment and follow-up
* Be willing to provide at least one collateral contact and collateral contact information

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 203 (Actual)
Dates: Start 2003-03; Primary Completion 2005-03 (Actual); Study Completion 2005-03 (Actual)

PRIMARY OUTCOMES:
Smoking Behavior
Smoking Cessation
Substance Abuse

CONTACTS AND LOCATIONS:
Overall Officials: Stephen F Butler, Ph.D., Principal Investigator — Inflexxion, Inc.
Locations (7):
- United States (7):
  - SPIRITT Family Services, La Puente, California
  - Athol Behavioral Health Center, Athol, Massachusetts
  - Home of New Vision, Ann Arbor, Michigan
  - New Life Home for Recovering Women, Inc, Detroit, Michigan
  - Brooklyn Psychiatric Centers, Brooklyn, New York
  - North General Hospital, New York, New York
  - Maple Leaf Counseling, Inc., Montpelier, Vermont